CLINICAL TRIAL: NCT05926570
Title: Parathyroid Hormone Level and Growth in Pediatric Patients With ESRD on Regular Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sara Mabrouk Elghoul, Principal Investigator, Clinical Lecturer of Pediatric Nephrology, Tanta University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 36264PR295/8/23
Record Dates: First submitted 2023-06-07; First posted 2023-07-03 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Drug Effect
Keywords: cinacalcet; insulin like growth factor-1
MeSH Terms: interventions — Cinacalcet

STUDY DESIGN:
Intervention Model Description: evaluate the effect of cinacalcet on insulin like growth factor-1 in pediatric patients with ESRD on regular hemodialysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 35 children and adolescents with end stage renal disease on regular hemodialysis (Experimental): All children will receive cinacalcet in a dose of 30 mg/day taken with food for 3 months
  Interventions: Drug: Cinacalcet

INTERVENTIONS:
Drug: Cinacalcet — calcimimetic
  Other Names: Mimpara

SUMMARY:
Chronic kidney disease (CKD) is defined as either renal damage and/ or a glomerular filtration rate (GFR) below 60 mL/min/1.73 m2 for more than 3 months. End stage renal disease (ESRD) is defined as GFR below 15 mL/min/1.73 m2.

Secondary hyperparathyroidism (SHPT) is an insidious disease that develops early in the course of CKD and increase in severity as the GFR deteriorates. High serum levels of intact parathyroid hormone (iPTH) are known to cause high turnover bone disease, i.e. osteitis fibrosa and have also been reported to increase the mortality risk in patients undergoing hemodialysis (HD).

Standard therapy for SHPT includes dietary calcium supplementation, active vitamin D, and phosphate binders; however, these are often insufficient to allow patients to achieve their serum parathyroid hormone (PTH), calcium and calcium-phosphorus product (Ca × P) targets.

Recent preclinical studies have demonstrated that treatment with calcimimetics that increase the sensitivity of the calcium-sensing receptor (CaR) to calcium can reverse the alterations in CaR and vitamin D receptor expression and parathyroid cell proliferation that are associated with SHPT.

Calcimimetics such as cinacalect are positive allosteric modulators of the calcium-sensing receptor that increase its sensitivity by lowering the threshold for activation by extracellular calcium ions. The calcimimetic cinacalcet mainly increases the sensitivity of the CaR to extracellular Ca, thus inhibiting the release of PTH, although, as recently shown, it also decreases PTH synthesis.

Growth hormone (GH) indirectly promotes the growth of child by stimulating the production of insulin like growth factor (IGF-1), many children with renal disease have normal or elevated level of GH in their blood otherwise the levels of IGF-1 are low because the approximately 98% of IGF-1 is always bound to one of binding proteins (BP) inside the liver, so this accumulated protein will reduce the function of IGF-1.

Using cinacalcet in controlling hyperparathyroidism may reduce growth problems in children with ESRD with regular hemodialysis.

DETAILED DESCRIPTION:
This interventional study will be conducted at Nephrology Unit Pediatric Department Tanta University Hospital (TUH) for a period of 6 months starting from August 2023.

Study duration 6 months from August 2023 to February 2024. Place of the study: Nephrology Unit at TUH. Study sample: This study will be conducted on 35 children and adolescents with end stage renal disease on regular hemodialysis for three to four times weekly at our nephrology Unit at TUH during the period of the study.

Inclusion criteria:

Pediatric patients with end stage renal disease aged from 8 to 18 years on regular hemodialysis.

Exclusion criteria:

* Controlled hyperparathyroidism- PTH <300 pg/ml.
* Children < 8y.
* Previous parathyroidectomy
* children on growth hormone therapy

All patients included in the study will be subjected to:

1. History taking including duration of dialysis and regular drugs that are taken.
2. Clinical examination including anthropometric measurements and blood pressure estimation. All measurements will be taken in the dialysis free day
3. Investigations A- Routine investigations: including

   * Complete blood picture
   * Serum albumin Serum creatinine, blood urea level●
   * Serum CRP B- Specific investigations: including

     * Serum insulin growth factor-1 using ELIZA kits.
     * Serum parathyroid hormone.
     * Serum calcium.
     * Serum phosphorus.
     * Serum alkaline phosphatase.

   Sample collection:

   Seven millilitres of venous blood will be collected under complete aseptic precautions at 8 AM and before dialysis session before and after one month of cinacalcet treatment. Five millilitres will be put in a plain test tube without anticoagulant, and the remaining two millilitres will be put in a test tube with ethylene diamine tetra-acetic acid (EDTA) as an anticoagulant, to be used for performing complete blood count. After clotting, the samples will be centrifuged at 1500 xg for 15 minutes. Part of the separated serum will be used to perform serum creatinine, urea, albumin and blood urea nitrogen (BUN). The rest of the serum will be separated and will be used for the subsequent assay of IGF-1 serum level by enzyme-linked immunosorbent assay (ELISA). Hemolysed samples will be discarded. Repeated thawing and freezing will be avoided.
4. treatment received: All children will receive cinacalcet in a dose of 30 mg/day taken with food for 3 months, in addition to their supportive treatment including erythropoietin injection, oral calcium, one alpha, folic acid and antihypertensive drugs to hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with end stage renal disease aged from 5 to 18 years on regular hemodialysis.

Exclusion Criteria:

* Controlled hyperparathyroidism- PTH <300 pg/ml.
* Children < 8y.
* Previous parathyroidectomy
* children on growth hormone therapy

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2023-08-05 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
correlation between PTH and serum IGF-1 | 3 months
  correlation between serum levels of parathyroid hormone and serum insulin like growth factor-1 in pediatric patients with ESRD on regular hemodialysis

SECONDARY OUTCOMES:
Cinacalcet effect on level of IGF-1 | 3 months
  cinacalcet will be given in a dose of 39mg/day with food for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sara Mabrouk Mohamed Elghoul, MD, Principal Investigator — Tanta University
Locations (1):
- Sara Mabrouk Mohamed Elghoul, Tanta, Egypt